CLINICAL TRIAL: NCT04275167
Title: Capsule Endomicroscopy for Visualization of the Small Intestine in EED Population in Pakistan
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Aga Khan University Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Guillermo Tearney, Guillermo J. Tearney, MD, PhD - Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2017P001219
Record Dates: First submitted 2019-12-09; First posted 2020-02-19 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Environmental Enteric Dysfunction
Keywords: Tethered Capsule Endomicroscopy; Optical Coherence Tomography; EED; Pakistan; Intestinal Disorder
MeSH Terms: conditions — Intestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Feasibility of TCE (Experimental): Feasibility is measured by the number of participants that we have successfully deployed the Tethered capsule device in.
  Interventions: Device: Tethered Capsule Endomicroscope/Trans Nasal Endomicroscope
- Feasibility of TNE and Microbiome Brushing (Experimental): Feasibility is measured by the number of participants that we have successfully deployed the TNE device and collected brush samples in.
  Interventions: Device: Tethered Capsule Endomicroscope/Trans Nasal Endomicroscope

INTERVENTIONS:
Device: Tethered Capsule Endomicroscope/Trans Nasal Endomicroscope — Either the Tethered Capsule Endomicroscope or the Transnasal Endomicroscope will be deployed in the subject. Once the capsule is swallowed /TNE device is inserted, the device will naturally be moved to the duodenum via peristalsis. Once in the duodenum, imaging will be performed. For subjects receiving the TNE device, brushing samples will be collected through the introduction tube.

SUMMARY:
This pilot study will test the feasibility and tolerability of the tethered OCT capsule and Trans Nasal Endomicroscopy probe and accessory devices for imaging the small intestine in subjects with EED and a matched non-EED cohort. This study will assess subject tolerability, optimal imaging technique, and imaging of EED features.

DETAILED DESCRIPTION:
Environmental enteric dysfunction (EED) is a poorly understood condition characterized by intestinal inflammation and loss of barrier function that is prevalent in regions of the world with inadequate sanitation and hygiene. EED is a major driver of malnourishment, poor neurological development, stunting, oral vaccine failure, and infection, affecting 25% of all children globally and causing over a million deaths each year . It is hypothesized that the stunting associated with EED begins in utero and that the mother's gut health has a significant impact on the fetus. Key periods of growth from pregnancy through birth and childhood offer windows for potential intervention Progress towards understanding EED and developing effective interventions has been hampered by an inability to evaluate the intestinal mucosa of populations in impoverished regions of the world where this condition is endemic.

The Tearney Laboratory has developed a minimally invasive screening method known as tethered capsule endomicroscopy (TCE) for imaging intestinal mucosa. With TCE, an unsedated subject swallows a tethered pill, which captures microscopic images of the entire esophagus, stomach, and small intestine, as it is naturally transits these organs via peristalsis and under the influence of gravity. The capsule implements a microscopic imaging technology called optical coherence tomography (OCT) that obtains 10-µm-resolution cross-sectional images of tissue. The procedure is brief, well tolerated, and can be much less expensive than endoscopy. The Investigators have implemented TCE for imaging the upper gastrointestinal tract of adults and adolescents with Celiac Disease (CD) and eosinophilic esophagitis (EoE), inflammatory conditions that are common in the US. The qualities seen thus far in their TCE studies - high imaging resolution, comprehensive tissue assessment, and minimal invasiveness - are also the qualities needed for evaluating the intestinal mucosa in populations with EED.

The Tearney Lab has also developed a new technique of deployment, Trans Nasal Endomicroscopy (TNE). The TNE catheter comprises of an introduction tube, similar to a standard Nasojejunal tube, with one or two balloons attached at the distal end. These balloons are inflated with Galinstan , a safe liquid metal alloy used in pediatric thermometers, or saline or sugar water or air which provides weight for the device to move to the duodenum under the forces of gravity and peristalsis. The TNE catheter encloses the OCT optics within, and is designed to have many of the same imaging properties of TCE but is introduced Trans nasally so that it can be effectively used in children, infants and also enable collection of various tissue samples using accessory probes for analysis through the lumen of the introduction tube.

There have been theories proposed that increased microorganism load and/or dysbiosis or an imbalance in the composition of gut microorganisms in the intestine may be important in the establishment and/or maintenance of EED. Duodenal Aspiration during endoscopy is currently used as gold standard for standard of care to collect targeted microbiome. However, the microbiome yield from this procedure is low and the procedure requires an EGD, which is a fairly invasive procedure, and carries all of the risks associated with an EGD . Tearney lab has developed a brush that can collect microbiota samples from the small intestine, in the unsedated subject in a non-invasive manner. The brush is similar to cytology brush used in standard clinical care, designed to be deployed through the TNIT tube.

The first phase of this study will test the feasibility and tolerability of the TCE device for imaging subjects with EED. The second phase of this study will test the TNE device and its accessories for imaging and microbial sample collection in pregnant women.

ELIGIBILITY:
The Inclusion Criteria:

* Children must be 6 months to 59 months old
* Adult participants 18 years of age or older scheduled for a standard of care endoscopy
* EED manifesting as malnourishment (WHZ<-2) without clear etiology or healthy subjects with WHZ >=0
* Participants and/or parents/guardians must be able to give informed consent/assent
* Participants and/or parents/guardians must be willing to provide consent for live streaming of the procedure
* Participants must be able to follow fasting instructions prior to the procedure

Inclusion criteria for Pregnant women:

* Participants 18 years and older
* Participants who are in their 2nd trimester of singleton pregnancy as confirmed by an ultrasound
* Participants with a BMI below 18.5 without clear etiology and healthy pregnant women with BMI between 18.5 -24.5.
* Participants must be able to follow fasting instructions prior to the procedure
* Participants must be able to consent to the procedure

Tethered Capsule Exclusion Criteria:

* Participants with any history of esophageal or intestinal strictures or prior GI surgery
* Participants with history of pyloric stenosis
* Participants with HIV diagnosis

Trans Nasal Exclusion Criteria:

* Participants with any contraindications for NG/NJ tube placement, including but not limited to those listed below:
* Participants with any history of esophageal or intestinal strictures or prior GI surgery
* Participants with history of pyloric stenosis or atresia
* Participants with suspected or diagnosed HIV, Hepatitis B and C
* Participants with any history of esophageal or intestinal strictures or prior GI surgery
* Participants with a history of upper gastrointestinal surgery including fundoplication
* Participants with upper GI obstruction
* Participants with short bowel syndrome
* Participants with upper respiratory infection at least 7 days prior to the procedure
* Deviated septum or any other anatomical abnormalities of the nasopharynx or upper gastrointestinal region, history of trans-sphenoidal surgery, facial or cranial trauma and fractures, chronic sinusitis, esophageal strictures, varices etc.
* Participants on drugs which impair clotting like anticoagulants and antiplatelet drugs, NSAIDS, history of bleeding disorders.
* Participants with upper GI bleeding

Microbiome Brush Exclusion Criteria

- Participants with any contraindications to gastrointestinal biopsies as per standard of care

For pregnant participants:

* Participants with high-risk pregnancy conditions at the discretion of the subject's physician and the PI
* Pregnant participants with a history of hyperemesis gravidarum
* Pregnant participants with a history of severe anemia
* Pregnant participants with gestational thrombocytopenia
* Pregnant participants with Type 1 diabetes
* Pregnant participants with Type 2 diabetes on medication and gestational diabetes requiring medication

Ages: 6 Months to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2017-10-11 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of TCE and TNE | up to 3 hours during the study.
  Number of participants that we have successfully deployed the Trans-nasal imaging device/Tethered capsule device in.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Tearney, M.D, PhD., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Aga Khan Medical Center, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: No